CLINICAL TRIAL: NCT03465787
Title: A Phase 3 Randomized, Double-Blind, Active-controlled Study to Evaluate the Efficacy and Safety of Lurasidone in Acutely Psychotic Patients With Schizophrenia
Brief Title: A 6-week Study to Evaluate the Efficacy and Safety of Lurasidone HCL in Acutely Psychotic Patients With Schizophrenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bukwang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BK-LuD-301
Record Dates: First submitted 2018-03-08; First posted 2018-03-14 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Acutely Psychotic Patients with Schizophrenia; Latuda; Lurasidone
MeSH Terms: conditions — Schizophrenia | interventions — Lurasidone Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lurasidone HCL 160 mg (Experimental): Lurasidone HCL 160 mg/day
  Interventions: Drug: Lurasidone HCL 160 mg
- Quetiapine XR 600 mg (Active Comparator): Quetiapine XR 600 mg/day
  Interventions: Drug: Quetiapine XR 600 mg

INTERVENTIONS:
Drug: Lurasidone HCL 160 mg — Lurasidone HCL 2 80mg tablets, QD
  Arms: Lurasidone HCL 160 mg
Drug: Quetiapine XR 600 mg — Quetiapine XR 2 300 mg tablets, QD
  Arms: Quetiapine XR 600 mg

SUMMARY:
This is a study designed to evaluate the efficacy and safety of lurasidone in acutely psychotic patients with chronic schizophrenia and to confirm the non-inferiority of lurasidone relative to quetiapine XR.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent and aged between 19 and 75 years of age.
2. Meets DSM-5 criteria for a primary diagnosis of schizophrenia.
3. CGI-S ≥ 4 at screening and baseline.
4. Subject is not pregnant (must have a negative serum pregnancy test at screening) or nursing (must not be lactating) and is not planning pregnancy within the projected duration of the study.
5. Subject is able and agrees to remain off prior antipsychotic medication for the duration of the study.
6. Subject is in good physical health on the basis of medical history, physical examination, and laboratory screening.

Exclusion Criteria:

1. The subject has evidence of any chronic organic disease of the CNS (other than schizophrenia)
2. Subject has participated in a prior trial of lurasidone.
3. Clinically significant or history of alcohol abuse/alcoholism or drug abuse/dependence within the last 6 months.
4. In the opinion of the investigator, subject is unable to cooperate with any study procedures, unlikely to adhere to the study procedures, keep appointments, or is planning to relocate during the study.
5. Considered by the investigator to be at imminent risk of suicide or injury to self, others, or property.

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2018-04-09 (Actual); Primary Completion 2022-10-26 (Actual); Study Completion 2022-10-26 (Actual)

PRIMARY OUTCOMES:
Mean change in Total PANSS Score From Baseline at Week 6 | Week 6
  The PANSS (Positive and Negative Syndrome Scale) is a 30-item scale (range 30-210) designed to assess various symptoms of schizophrenia including delusions, grandiosity, blunted affect, poor attention, and poor impulse control. The 30 symptoms are rated on a 7-point scale that ranges from 1 (absent) to 7 (extreme psychopathology). The PANSS total score consists of the sum of all 30 PANSS items. Higher scores indicate worsening.

SECONDARY OUTCOMES:
Mean change in CGI-S score From Baseline at Week 6 | Week 6
  Clinical Global Impression of Severity is a clinician-rated assessment of the subject's current illness state on a 7 point scale, where a higher score is associated with greater illness severity. The scale has a single item measured on a 7 point scale from 1 ('normal', not ill) to 7 (extremely ill).

CONTACTS AND LOCATIONS:
Overall Officials: Jung Hee Yeon, Principal Investigator — SMG-SNU Boramae Medical Center
Locations (1):
- Borame Medical Center, Seoul, Seoul, Dongjak-gu, South Korea